CLINICAL TRIAL: NCT03055832
Title: Randomized Comparison Between iLux™ and LipiFlow® in the Treatment of Meibomian Gland Dysfunction
Brief Title: Comparison Between iLux™ and LipiFlow® in the Treatment of Meibomian Gland Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tear Film Innovations, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-03
Record Dates: First submitted 2017-02-10; First posted 2017-02-16 (Actual); Results first posted 2019-05-20 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2019-05

CONDITIONS: Meibomian Gland Dysfunction
Keywords: iLux; LipiFlow; dry eye; Meibomian Gland Dysfunction; evaporative dry eye
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Meibomian gland score will be assessed by a masked rater
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- iLux 2020 System (Experimental): Meibomian gland treatment (Day 0) according to instructions for use (IFU)/User Manual
  Interventions: Device: iLux 2020 System
- LipiFlow Thermal Pulsation System (Active Comparator): Meibomian gland treatment (Day 0) according to instructions for use (IFU)/User Manual
  Interventions: Device: LipiFlow Pulsation System

INTERVENTIONS:
Device: iLux 2020 System — Medical device that applies localized heat and pressure therapy to the eyelid in order to express melted meibum from obstructed glands
  Arms: iLux 2020 System
Device: LipiFlow Pulsation System — Medical device that applies a combination of heat and pressure to the inner eyelid to remove gland obstructions and stagnant gland content
  Arms: LipiFlow Thermal Pulsation System

SUMMARY:
The purpose of this study was to compare changes in meibomian gland dysfunction (MGD), tear break-up time (TBT) and evaporative dry eye (EDE) symptoms after treatment with either the iLux® 2020 System or the LipiFlow® Thermal Pulsation System.

DETAILED DESCRIPTION:
At the Baseline visit (Day 0), subjects were assessed pre-treatment, during treatment, and post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older of any gender or race
* Written informed consent to participate in the study
* Willingness and ability to return for all study visits
* Positive history of self-reported dry eye symptoms for three months prior to the study using OSDI with a score of ≥ 23 at the baseline visit
* Evidence of meibomian gland (MG) obstruction, based on total MGS of ≤12 in lower eyelids for each eye as assessed by a clinician not involved in the study procedure
* Tear break-up time <10 seconds
* Agreement/ability to abstain from dry eye/MGD medications for the time between the screening visit and the final study visit (ocular lubricants are allowed if no changes are made during the study)

Exclusion Criteria:

* History of ocular or corneal surgery including intraocular, oculo-plastic, corneal or refractive surgery within 1 year
* Subjects with giant papillary conjunctivitis
* Subject with punctal plugs or who have had punctal cautery
* Ocular injury or trauma, chemical burns, or limbal stem cell deficiency within 3 months of the baseline examination
* Active ocular herpes zoster or simplex of eye or eyelid or a history of these within the last 3 months
* Subjects who are aphakic
* Cicatricial lid margin disease identified via slit lamp examination, including pemphigoid, symblepharon, etc.
* Active ocular infection
* Active ocular inflammation or history of chronic, recurrent ocular inflammation within prior 3 months
* Ocular surface abnormality that may compromise corneal integrity
* Lid surface abnormalities that affect lid function in either eye
* Anterior blepharitis (staphylococcal, demodex or seborrheic grade 3 or 4)
* Systemic disease conditions that cause dry eye
* Unwillingness to abstain from systemic medications known to cause dryness for the study duration
* Women who are pregnant, nursing, or not utilizing adequate birth control measures
* Individuals who have either changed the dosing of systemic medications or non-dry eye/MGD ophthalmic medications within the past 30 days prior to screening
* Individuals who are unable or unwilling to remain on a stable dosing regimen for the duration of the study
* Individuals using isotretinoin (Accutane) within 1 year, cyclosporine-A (Restasis) or lifitegrast ophthalmic solution 5% (Xiidra) within 3 months, or any other dry eye or MGD medications within 2 weeks of screening (ocular lubricants are allowed if no changes are made during the study)
* Individuals wearing contact lenses at any time during the prior three months or during the study period
* Eyelid tattoos, including permanent eyeliner makeup
* Individuals that were treated with LipiFlow in either eye in the last 24 months
* Individuals using another ophthalmic investigational device or agent within 30 days of study participation
* Individuals who are unable to complete the required patient questionnaires in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-07-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - TearFilm Investigative Site, Phoenix, Arizona
  - TearFilm Investigative Site, Scottsdale, Arizona
  - TearFilm Investigative Site, San Diego, California
  - TearFilm Investigative Site, Centennial, Colorado
  - TearFilm Investigative Site, Greenwood Village, Colorado
  - TearFilm Investigative Site, Chesterfield, Missouri
  - TearFilm Investigative Site, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Baseline
Arm/Group | iLux 2020 System | LipiFlow Thermal Pulsation System
Started | 71 | 71
Completed | 71 | 71
Not Completed | 0 | 0
Period: Immediately Post-Procedure (Hour 1)
Arm/Group | iLux 2020 System | LipiFlow Thermal Pulsation System
Started | 71 | 71
Completed | 71 | 71
Not Completed | 0 | 0
Period: Day 1
Arm/Group | iLux 2020 System | LipiFlow Thermal Pulsation System
Started | 71 | 71
Completed | 71 | 71
Not Completed | 0 | 0
Period: Week 2
Arm/Group | iLux 2020 System | LipiFlow Thermal Pulsation System
Started | 71 | 71
Completed | 70 | 71
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Week 4
Arm/Group | iLux 2020 System | LipiFlow Thermal Pulsation System
Started | 70 | 71
Completed | 70 | 71
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | iLux 2020 System | LipiFlow Thermal Pulsation System | Total
Number analyzed (Participants) | 71 | 71 | 142
Age, Customized [Count of Participants; unit: Participants]
  Under 18 Years | 0 | 0 | 0
  18 Years and Older | 71 | 71 | 142
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 49 | 101
  Male | 19 | 22 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 61 | 68 | 129
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 71 | 71 | 142

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 4 in Meibomian Gland Score (MGS)
Description: Meibomian glands on the lower eyelid were assessed by the examiner using a Meibomian Gland Evaluator while viewing the eyelid margin using a slit lamp microscope. 5 glands in 3 zones (nasal, medial, temporal) were evaluated. Each gland was scored from 0-3 for a maximum MGS of 45 in each eye. MGS scoring was as follows: 0 = no secretion (worst), 1 = inspissated, 2 = cloudy, 3 = clear liquid (best). A positive change value indicates an improvement.
Time Frame: Baseline, Week 4
Population: All randomized and treated patients
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Groups:
- iLux Right Eye: Right Eye of Subjects treated with the iLux 2020 System
- iLux Left Eye: Left Eye of Subjects treated with the iLux 2020 System
- iLux Both Eyes: Both Eyes of Subjects treated with the iLux 2020 System
- LipiFlow Right Eye: Right Eye of Subjects Treated with the LipiFlow Thermal Pulsation System
- LipiFlow Left Eye: Left Eye of Subjects treated with Lipiflow Thermal Pulsation System
- LipiFlow Both Eyes: Both Eyes of Subjects treated with the LipiFlow Thermal Pulsation System
Arm/Group | iLux Right Eye | iLux Left Eye | iLux Both Eyes | LipiFlow Right Eye | LipiFlow Left Eye | LipiFlow Both Eyes
Number analyzed (Participants) | 70 | 70 | 70 | 70 | 71 | 71
Number analyzed (Eyes) | 70 | 70 | 140 | 70 | 71 | 141
score on a scale | 17.3 (12.1) | 18.0 (12.2) | 17.7 (12.2) | 18.1 (10.8) | 16.9 (11.5) | 17.5 (11.1)
Statistical Analysis 1: Comparison: iLux Both Eyes vs LipiFlow Both Eyes; Test type: Non-Inferiority — This study provides a combined power of co-primary endpoints of 88% given the following primary endpoint assumptions: * MGS non-inferiority delta of 5 points and standard deviation of 8 points provides power of 93.9% * TBT non-inferiority delta of 2.5 seconds and standard deviation of 4 seconds, provides a TBT primary endpoint power of 93.9% * Power that both endpoitns are significant, assuming independence was 0.939^2 = 0.882 or 88.2% power; Mean Difference (Net) = -0.13, 95% CI 2-sided [-3.82 to 3.56], Standard Error of Mean 1.88

2. Primary Outcome: Change From Baseline to Week 4 in Tear Break-Up Time (TBT)
Description: Tear break-up time (defined as the time required for dry spots to appear on the surface of the eye after blinking) was assessed by the examiner using a slit lamp and fluorescein strips. Fluorescein was instilled onto the patient's eye, after which the patient blinked three times, then kept the eye open. Immediately thereafter, the examiner used a stopwatch to record the time between the last blink and the first appearance of a dark spot on the cornea (formation of dry area). Three consecutive measurements were taken and averaged for actual TBT. A positive change value represents a lengthening in the tear break-up time and greater comfort.
Time Frame: Baseline, Week 4
Population: All randomized and treated patients
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: Eyes
Arm/Group | iLux Right Eye | iLux Left Eye | iLux Both Eyes | LipiFlow Right Eye | LipiFlow Left Eye | LipiFlow Both Eyes
Number analyzed (Participants) | 70 | 70 | 70 | 71 | 71 | 71
Number analyzed (Eyes) | 70 | 70 | 140 | 71 | 71 | 142
seconds | 2.86 (3.72) | 2.73 (3.72) | 2.79 (3.66) | 2.69 (3.31) | 2.61 (3.22) | 2.65 (3.25)
Statistical Analysis 1: Comparison: iLux Both Eyes vs LipiFlow Both Eyes; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.10, 95% CI 2-sided [-0.97 to 1.16], Standard Error of Mean 0.54

3. Primary Outcome: Incidence (Number) of Device- or Procedure-related Adverse Events
Description: The number of device- or procedure-related adverse events was calculated, including changes from baseline (Yes/No) in any of the following eyelid characteristics: lid margin assessment or development of floppy eyelids or entropion (eyelid rolled inward) or ectropion (eyelid sagging outward) or loss of lash integrity.
Time Frame: Week 4
Population: All randomized and treated patients
Measure: Number; unit: Adverse event
Groups:
- iLux 2020 System: Meibomian Gland Treatment
  iLux 2020 System: Heating and compression to express clogged meibomian glands
- LipiFlow Thermal Pulsation System: Meibomian Gland Treatment
  LipiFlow Pulsation System: Heating and compression to express clogged meibomian glands
Arm/Group | iLux 2020 System | LipiFlow Thermal Pulsation System
Number analyzed (Participants) | 70 | 71
Adverse event | 4 | 0
Statistical Analysis 1: Comparison: iLux 2020 System vs LipiFlow Thermal Pulsation System; Test type: Other — A formal hypothesis was not proposed for this endpoint and therefore a power calculation was not performed. A Fisher's Exact test was performed post hoc to determine if a significant difference existed between the two arms; p = 0.12, Fisher Exact

4. Secondary Outcome: Change From Baseline to Week 4 in Ocular Surface Disease Index (OSDI)
Description: The Ocular Surface Disease Index (OSDI) is a 12-item, patient-reported outcome questionnaire used to measure ocular symptoms, visual function, and environmental factors that may affect a patient's vision. Each item is scored on a 0-4 Likert-type scale, where 0 is "None" and 4 is "All of the Time." The OSDI is calculated as the (sum of scores) x 25 / (# of questions answered), for a resultant overall score of 0-100, where 0 corresponds to no disability and 100 corresponds to complete disability. A negative change value indicates an improvement.
Time Frame: Baseline, Week 4
Population: All randomized and treated patients
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- iLux All Questions: All OSDI questions in Subjects treated with the iLux 2020 System
- iLux Vision Questions: OSDI Questions 1-5 in Subjects Treated with the iLux 2020 System
- iLux Ocular Questions: OSDI questions 6-9 in Subjects treated with the iLux 2020 System
- iLux Trigger Questions: OSDI questions 10-12 in Subjects treated with the iLux 2020 System
- LipiFlow All Questions: All OSDI questions (1-12) in Subjects treated with the LipiFlow Thermal Pulsation System
- LipiFlow Vision Questions: OSDI Questions 1-5 in Subjects treated with the LipiFlow Thermal Pulsation System
- LipiFlow Ocular Questions: OSDI questions 6-9 in Subjects treated with the LipiFlow Thermal Pulsation System
- LipiFlow Trigger Questions: OSDI questions 10-12 in Subjects treated with the LipiFlow Thermal Pulsation System
Arm/Group | iLux All Questions | iLux Vision Questions | iLux Ocular Questions | iLux Trigger Questions | LipiFlow All Questions | LipiFlow Vision Questions | LipiFlow Ocular Questions | LipiFlow Trigger Questions
Number analyzed (Participants) | 70 | 70 | 70 | 70 | 71 | 71 | 70 | 71
score on a scale | -31.0 (18.4) | -27.3 (19.7) | -30.9 (25.9) | -37.0 (30.6) | -28.0 (22.8) | -24.9 (20.0) | -27.5 (28.4) | -34.4 (34.7)
Statistical Analysis 1: Comparison: iLux All Questions vs LipiFlow All Questions; All questions; Test type: Non-Inferiority — A standard deviation of 14 was assumed based on pilot data and the non-inferiority delta was set to 7. The chosen sample size and alpha = 0.025 provides 80% power for this endpoint; Mean Difference (Net) = -3.08, 95% CI 2-sided [-8.75 to 2.59], Standard Error of Mean 2.89

5. Secondary Outcome: Mean Pain Score During Treatment
Description: The patient placed a vertical line on visual analog scale questionnaire using a scale of 0-100 (0 = no pain, 100 = maximum pain) at the point that indicated the pain in or around their eyelids, or face during the procedure including feelings of pressure, tightness, heaviness, burning, and other negative sensations. A score a 20 was associated with a description of "hurts a little". Assessments were made at baseline (pre-treatment), immediately post-treatment, and Day 1 post-treatment. No formal hypothesis testing was pre-specified for this endpoint.
Time Frame: Baseline (Day 0), Immediately Post-Treatment (Day 0), Day 1 Post-Treatment
Population: All randomized and treated patients
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | iLux Right Eye | iLux Left Eye | iLux Both Eyes | LipiFlow Right Eye | LipiFlow Left Eye | LipiFlow Both Eyes
Number analyzed (Participants) | 71 | 71 | 71 | 69 | 70 | 70
Number analyzed (Eyes) | 71 | 71 | 142 | 69 | 70 | 139
score on a scale
  Baseline (Day 0) | 34.4 (28.6) | 34.0 (28.0) | 34.2 (28.2) | 30.8 (26.4) | 32.6 (27.6) | 31.7 (27.0)
  Immediately Post-Treatment (Day 0) | 25.2 (25.1) | 23.6 (23.7) | 24.4 (24.3) | 10.2 (14.6) | 10.1 (13.8) | 10.1 (14.1)
  Day 1 Post-Treatment | 12.0 (15.7) | 13.0 (17.0) | 12.5 (16.3) | 11.8 (17.8) | 11.5 (16.9) | 11.7 (17.3)

6. Secondary Outcome: Mean Discomfort Score During Treatment
Description: The patient placed a vertical line on visual analog scale questionnaire using a scale of 0-100 (0 = no discomfort, 100 = maximum discomfort) at the point that indicated the discomfort in or around their eyelids, or face during the procedure including feelings of pressure, tightness, heaviness, burning, and other negative sensations. Assessments were made at baseline (pre-treatment), immediately post-treatment, and Day 1 post-treatment. No formal hypothesis testing was pre-specified for this endpoint.
Time Frame: Baseline (Day 0), Immediately Post-Treatment (Day 0), Day 1 Post-Treatment
Population: All randomized and treated patients
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | iLux Right Eye | iLux Left Eye | iLux Both Eyes | LipiFlow Right Eye | LipiFlow Left Eye | LipiFlow Both Eyes
Number analyzed (Participants) | 71 | 71 | 71 | 69 | 70 | 70
Number analyzed (Eyes) | 71 | 71 | 142 | 69 | 70 | 139
score on a scale
  Baseline (Day 0) | 56.3 (22.3) | 55.9 (21.8) | 56.1 (22.0) | 52.1 (23.6) | 52.6 (24.0) | 52.3 (23.6)
  Immediately Post-Treatment (Day 0) | 38.9 (24.7) | 36.7 (22.5) | 37.8 (23.6) | 22.3 (21.2) | 23.7 (21.6) | 23.0 (21.3)
  Day 1 Post-Treatment | 23.5 (22.5) | 23.7 (22.4) | 23.6 (22.4) | 24.7 (24.2) | 24.4 (23.4) | 24.5 (23.7)

7. Secondary Outcome: Change From Baseline to Post-Treatment in Ocular Surface Staining
Description: Corneal staining was assessed by the examiner using the National Eye Institute corneal grading scale and a slit-lamp. Each of the 5 corneal regions (superior, inferior, central, temporal, & central), was graded on a 0-3 scale, where 0=normal-no staining (best); 1=mild-superficial stippling micropunctate staining; 2=moderate-macropunctate staining with some coalescent areas; and 3=severe-numerous coalescent macropunctate areas and/or patches (worst). The scores were summed for each eye, and an overall corneal staining score was computed as the average of the sum from both eyes. Overall scores ranged between 0-15, with higher change value indicating greater damage to the corneal surface. Assessments were made at baseline (pre-treatment), immediately post-treatment, and Day 1 post-treatment. No formal hypothesis testing was pre-specified for this endpoint.
Time Frame: Baseline (Day 0), Immediately Post-Treatment (Day 0), Day 1 Post-Treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | iLux Right Eye | iLux Left Eye | iLux Both Eyes | LipiFlow Right Eye | LipiFlow Left Eye | LipiFlow Both Eyes
Number analyzed (Participants) | 71 | 71 | 71 | 70 | 70 | 70
Number analyzed (Eyes) | 71 | 71 | 142 | 70 | 70 | 140
score on a scale
  Change from Baseline to Immediately Post-Treatment | 0.6 (1.7) | 0.6 (1.7) | 0.6 (1.7) | 0.5 (1.6) | 0.4 (1.5) | 0.4 (1.6)
  Change from Baseline to Day 1 Post-Treatment | -0.9 (1.8) | -1.0 (2.0) | -0.9 (1.9) | -0.9 (1.5) | -1.2 (1.9) | -1.1 (1.7)

8. Secondary Outcome: Change From Baseline to Post-Treatment in Intraocular Pressure (IOP)
Description: IOP (fluid pressure inside the eye) was measured by Goldmann applanation tonometry. A higher IOP can be a greater risk for developing glaucoma or glaucoma progression (leading to optic nerve damage). A negative change value indicates an improvement. No formal hypothesis testing was pre-specified for this endpoint.
Time Frame: Baseline (Day 0), Immediately Post-Treatment (Day 0)
Population: All randomized and treated patients
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: Eyes
Arm/Group | iLux Right Eye | iLux Left Eye | iLux Both Eyes | LipiFlow Right Eye | LipiFlow Left Eye | LipiFlow Both Eyes
Number analyzed (Participants) | 71 | 71 | 71 | 69 | 69 | 69
Number analyzed (Eyes) | 71 | 71 | 142 | 69 | 69 | 138
mmHg | 0.04 (1.44) | -0.07 (1.54) | -0.01 (1.49) | 0.07 (1.94) | -0.04 (1.79) | 0.01 (1.86)

9. Secondary Outcome: Change From Baseline to Post-Treatment in Best Spectacle-Corrected Visual Acuity (BSCVA)
Description: Visual acuity was assessed with spectacles or other visual corrective devices in place using Early Treatment Diabetic Retinopathy Study (ETDRS) charts. Results are presented in logarithm of the minimum angle of resolution (logMAR) with 0.2 in logMAR corresponding to 10 ETDRS letters read. A lower logMAR change value indicates an improvement in visual acuity. No formal hypothesis testing was pre-specified for this endpoint.
Time Frame: Baseline (Day 0), Immediately Post-Treatment (Day 0)
Population: All randomized and treated patients
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | iLux Right Eye | iLux Left Eye | iLux Both Eyes | LipiFlow Right Eye | LipiFlow Left Eye | LipiFlow Both Eyes
Number analyzed (Participants) | 71 | 71 | 71 | 70 | 70 | 70
Number analyzed (Eyes) | 71 | 71 | 142 | 70 | 70 | 140
logMAR | 0.02 (0.08) | 0.05 (0.11) | 0.03 (0.09) | 0.02 (0.11) | 0.02 (0.07) | 0.02 (0.09)

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: Any untoward and unintended sign, symptom or disease temporally associated with the use of an investigational drug or device, or other protocol-imposed intervention, regardless of the suspected cause. Chronic but stable conditions or diseases are not AEs. Changes in a chronic condition or disease consistent with natural disease progression are not AEs. AEs were assessed during procedure, immediately post-procedure, 1 day, 2 weeks, & 4 weeks post-procedure.
Arm/Group | iLux 2020 System | LipiFlow Thermal Pulsation System
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/71
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/71
Other Adverse Events (participants affected / at risk) | 5/71 | 4/71
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iLux 2020 System (N=71) | LipiFlow Thermal Pulsation System (N=71)
Other (Eye disorders) | 5 (5) | 4 (4) — Includes: burning sensation, itching, stinging, petechial hemorrhage, superficial punctate keratitis, and blurred vision

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/32/NCT03055832/Prot_SAP_000.pdf